CLINICAL TRIAL: NCT06858605
Title: The Effect of Neck Mobilization vs. Combined Neck and Lumbar Mobilization on Pain and Range of Motion in People With Cervical Disc Herniation: A Randomized Controlled Study
Brief Title: Effect of Neck vs. Combined Neck-Lumbar Mobilization on Pain and Motion in Cervical Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Başar Öztürk, Assoc. Prof., Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: fztduygu
Record Dates: First submitted 2025-02-24; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Cervical Disc Herniation
Keywords: Intervertebral Disc Displacement; Musculoskeletal Manipulations; Range of Motion; Articular; Neck pain
MeSH Terms: conditions — Intervertebral Disc Displacement; Neck Pain

STUDY DESIGN:
Intervention Model Description: After obtaining informed consent forms from the participants who accepted to join the study, participants were randomly assigned to two groups-Group A (cervical-only KEOMT) and Group B (combined cervical and lumbar KEOMT)-using a computer-generated randomization sequence. Block randomization was employed to ensure balanced group sizes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Cervical mobilization group) (Experimental): Cervical mobilizations were performed with patients in a supine position. This setup facilitated accurate application of manual therapy techniques. Techniques included Grade 1 mobilizations (pain relief) and Grade 2 mobilizations (soft tissue relaxation). The concave-convex rule guided gliding and translatory movements for optimizing joint mechanics. Manual traction and segmental mobilization were performed with patients in a supine position. The KEOMT included cervical segmental traction and cervical segmental mobilization-flexion and gliding therapy in grade 3. The Convex/Concave Rule was consistently applied in all cases.
  Interventions: Other: Kaltenborn-Evjenth Orthopedic Manual Therapy (KEOMT)
- Group B (Combined cervical and lumbar mobilization group) (Experimental): For segmental flexion mobilization, the patient is positioned on their side with their hips and knees flexed. The therapist places one hand on the vertebrae, positioning the fingers on either the transverse or spinous processes, and the other hand on the sacrum in a similar manner. To facilitate movement, the therapist's chest makes contact with the patient's knees, allowing the pelvis to be guided in a caudal or ventral direction. This technique can be effectively adapted for both cervical and lumbar regions, maintaining consistent application across various spinal segments. For segmental traction, the patient also lies on their side, with their knees flexed toward the abdomen. The therapist hooks their fingers over the proximal transverse processes or the soft tissues in the paravertebral region and applies traction by pulling in opposite directions.
  Interventions: Other: Kaltenborn-Evjenth Orthopedic Manual Therapy (KEOMT)

INTERVENTIONS:
Other: Kaltenborn-Evjenth Orthopedic Manual Therapy (KEOMT) — Kaltenborn's biomechanical approach to diagnosis and treatment emphasizes ergonomic principles and trial-based techniques. His mobilization methods, classified into Grades I-III, target pain relief (Grades I-II) and joint hypomobility (Grade III) by enhancing glide and tissue elasticity. The Kaltenborn-Evjenth Orthopedic Manual Therapy (KEOMT) further refines this approach using arthrokinematic principles to restore physiological joint motion based on the concave-convex rule.

SUMMARY:
Background To assess the effectiveness of Kaltenborn-Evjenth Orthopedic Manual Therapy (KEOMT) applied to cervical-only mobilization versus both lumbar and cervical regions on pain intensity and range of motion (ROM) in individuals with cervical disc herniation, Methods: Thirty three participants were enrolled in the study. The patients were randomly assigned to two groups. Group A received cervical-only KEOMT while Group B received combined lumbar and cervical KEOMT, Interventions were administered three times a week for four weeks. Pain was measured using the Visual Analog Scale (VAS), ROM was assessed for flexion and lateral flexion, and Neck Pain and Disability Index (NPDI) and Short-Form 36 Health Survey (SF-36) were used for evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cervical disc herniation at least 8 weeks but not more than 5 years prior.
* Cervical disc herniation verified by magnetic resonance imaging (MRI) at 1 or 2 segmental levels, consistent with clinical findings.
* Neck Disability Index (NDI) score greater than 5.
* No use of analgesic medication other than the prescribed treatment before or during the study period.

Exclusion Criteria:

* History of myelopathy, whiplash-associated disorder, generalized myalgia, malignant tumor, or inflammatory disease.
* Painful back problems or neurological symptoms within the past year.
* Psychiatric disorders or drug abuse.
* Contraindications to physical therapy or inability to return to work or perform physical therapy due to other diseases or disabilities.
* Inability to communicate effectively.
* Participation in any additional interventions outside the prescribed treatment during the study period.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Visuel Analog Scale | Through study completion, an average of 1 year
  Pain intensity was evaluated with a visual analog scale (VAS). A 10 cm visual scale was divided into equal segments and numbered from 0 to 10. Patients were instructed that 0 represents no pain, while 10 indicates unbearable pain. Based on this explanation, they were asked to rate their pain intensity accordingly
Range of motion | Through study completion, an average of 1 year
  A universal goniometer was used to measure joint position and range of motion, following the guidelines of Kendall and the American Association of Orthopedic Surgeons. The assessment was conducted with the patient in a sitting position. Patients were instructed to actively perform movements of cervical flexion, extension, right and left rotation, and right and left lateral flexion, with the corresponding degrees of motion recorded.
Neck Pain and Disability Assessment | Through study completion, an average of 1 year
  Neck pain and disability were evaluated using the Neck Pain Disability Index (NPDI), a validated tool developed by Vernon and Mior (1991). The index comprises 20 items scored on a Visual Analog Scale (VAS), assessing the impact of neck pain on daily activities, occupational performance, and emotional well-being. Scores range from 0 (no disability) to 100 (complete disability), with higher scores indicating greater functional limitations. This study employed the Turkish version of the NPDI, which has demonstrated reliability
Quality of life scale | Through study completion, an average of 1 year
  The participants' quality of life was assessed using the Short Form 36 (SF-36), a self-reported scale developed by the Rand Corporation in 1992. The SF-36 evaluates general health status through 36 questions, divided into 8 subscales: physical function, physical role limitations, bodily pain, general health, vitality, social function, emotional well-being, and mental health. Scores on the SF-36 range from 0 to 100, with 0 representing the worst health status and 100 representing the best. The Turkish version of the scale was used in this study

CONTACTS AND LOCATIONS:
Locations (1):
- Fenerbahçe University Faculty of Health Sciences Physiotherapy Department, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ozdincler A, Aktas D, Aktar Reyhanioglu D, Ozturk B. The effect of neck mobilization Vs. combined neck and lumbar mobilization on pain and range of motion in people with cervical disc herniation: A randomized controlled study. J Bodyw Mov Ther. 2025 Sep;43:188-195. doi: 10.1016/j.jbmt.2025.04.032. Epub 2025 Apr 26. PMID 40483122